

# L'aîné au cœur de son milieu de vie - Social participation and community spirit in retirement homes

Presented to the Véritas IRB Research Ethics Committee

**TOPMED** 

**Version 01** 

Date: January 2024



# RESEARCH PROJECT DESCRIPTION SCHEDULED START AND END DATES

January 2024 to December

#### **PROJECT TITLE**

RD-23\_0437\_L'aîné au cœur de son milieu de vie - Social participation and community spirit in retirement homes

#### **QUALITIES AND SKILLS OF RESEARCH TEAM MEMBERS**

### **Principal Investigator**

Édith Martin, Ph.D., Director - Research and Innovation TOPMED CCTT, Collège Mérici 755 Grande-Allée West, Quebec City, Qc, G1S 1C1 (418) 683-2104, ext. 1302 emartin@topmed.ca

# Relevant experience

TOPMED researcher since 2014
B.Ing. Metallurgical Engineering (Materials orientation)
M.Sc.A. Biomedical Engineering
Ph.D. Metallurgical Engineering

# **Project coordinator**

Estelle Houguet
Research professional
TOPMED CCTT, Collège Mérici
755 Grande-Allée West, Quebec City, Qc, G1S 1C1
(418) 683-2104, ext. 1310
ehouguet@topmed.ca

Relevant experience M.Sc. Industrial Relations D.E.S.S Occupational Health and Safety

#### Other team members

Catherine Lavoie, T.P., Orthotist-Prosthetist, Research Professional TOPMED CCTT, Collège Mérici 755 Grande-Allée West, Quebec City, Qc, G1S 1C1 (418) 683-2104, ext. 1309 <a href="mailto:clavoie@topmed.ca">clavoie@topmed.ca</a>

Relevant experience (current position, qualifications)
DEC. Technique in orthotics and orthopaedic prosthetics



Mathieu Germain Robitaille, M.Sc. Kinesiologist, research professional TOPMED CCTT, Collège Mérici 755 Grande-Allée West, Quebec City, Qc, G1S 1C1 (418) 683-2104, ext. 1310 mgrobitaille@topmed.ca

Relevant experience (current position, qualifications)

B.Sc. Kinesiology M.Sc. Kinesiology

Céline Gagnon, M.Sc. teacher in the Special Education Techniques program Collège Mérici 755 Grande-Allée West, Quebec City, Qc, G1S 1C1 (418)683-1591 ext. 3323

20 years teaching special education techniques 14 years as a specialized educator for elderly clients with loss of autonomy (day center, CHSLD)

DEC Techniques en éducation spécialisée

Bacc. Multidisciplinary with specialization in gerontology

M.Sc Gérontologie- in progress

Isabelle Tremblay, Research Professional

TOPMED CCTT, Collège Mérici 755 Grande-Allée West, Quebec City, Qc, G1S 1C1 (418) 683-2104, ext. 1308 itremblay@topmed.ca

Relevant experience (current position, qualifications)
Certificate in sociology,
Participation in geronto-technology research projects,
Optimization of RPP sports facilities

#### **SOURCE OF FINANCING**

The project is funded by the French Ministry of Higher Education.

#### **PARTNER COMPANY**

SEC Fonds Immobilier Groupe John Conway, Consultant

Tel.: (514)

E-mail: JConway@legroupemaurice.com

#### RESEARCH PROJECT DESCRIPTION

#### Issues

Internationally, in Canada and in Quebec, the social participation (SP) of seniors is now at the heart of government issues. But social participation is not always easy. There are a number of factors that can influence its success. At a time when there are more and more places to live for the elderly, how can we offer optimal conditions for adequate



social participation for seniors? The links between participation and a sense of belonging are discussed in the literature. There are a few examples of structures that can help foster this feeling, such as the "Alzheimer homes" that are beginning to be set up in Europe and, more recently, in Canada. The question that arises, then, is how to envisage and enable the emergence of this sense of belonging, a fortiori in living environments such as retirement homes, where the elderly move around, often resulting in a loss of identity and landmarks.

Le Groupe Maurice is a Quebec-based group specializing in the design, development and management of residences for the elderly, which aims to embody the possibility of "better aging" by meeting the aspirations of seniors. With a view to offering the best possible services, including activities that foster optimal social participation, Groupe Maurice is now keen to understand and foster the conditions for social participation, notably through the emergence and sustainability of a sense of belonging and community spirit, particularly in the wake of the pandemic that has unfortunately forced seniors into physical and social isolation.

Building on multiple collaborations with TOPMED and Collège Mérici in applied research on enabling environments to promote mobility and autonomy, Groupe Maurice is now calling on the college and its CCTT to create a social innovation that will document the determinants of social participation (facilitators and obstacles) and highlight the challenges and possible solutions for fostering a sense of community in RPAs. Ultimately, Le Groupe Maurice would like to have a solution that can be transferred to all its seniors' facilities.

# State of knowledge and project relevance

Definition: Social participation (SP), understood as both a process and an outcome, can be defined as "taking part in activities of a social nature, i.e. maintaining meaningful relationships, being part of a community, and taking part in group activities, volunteering or paid work" (Public Health, 2018). Its definition, however, does not enjoy consensus within the literature.

Widely perceived as contributory, it can refer to the performance of daily activities, social interactions, integration into a social network or participation in a group of activities of a social nature recognized as being of public interest, such as associations (Raymond et al., 2008). However, this contributory acception could be overtaken when it comes to older people, as suggested by Raymond, Grenier and Hanley (2014), who highlight the need to understand social participation as "a reflection of the choices and needs of older people". Even so, having a unitary definition would facilitate study around the concept of "active aging" (Levasseur et al., 2022).

An important dimension of well-being for the elderly: The way we think about PS and its sustainability is all the more important since it has benefits for the elderly. From a health perspective, the literature highlights a positive and significant effect on "slowing cognitive and functional decline, reducing medication consumption, improving perception of health status and well-being" (Dadmar, Berrut & Campéon., 2018; Gilmour, 2012; Newman & Zainal, 2020; Raymond et al., 2008) as well as an impact on the risk of depression (Shiba et al., 2021). In addition, PS is recognized as a factor in combating social isolation, a way of increasing self-esteem and feelings of usefulness (Le Guen, 2001) or a way of increasing individual coping skills (Altintas et al, 2010; Dadmar, Berrut & Campéon, 2018). At the same time, studies recognize the benefit of SP at the collective level, since it can be a means of fostering a sense of belonging and attachment, where disabilities and limitations are often risks of social exclusion.

Determinants, facilitators and obstacles: The determinants of this participation need to be considered in the context of active ageing. In this respect, the literature distinguishes four categories of factors influencing PS. Socio-demographic factors, personal factors, environmental factors and social network factors. Socio-demographic factors include age, gender, education and marital status. In some cases, there also appears to be a socio-cultural and cross-cultural effect on social participation (Townsend et al., 2021). Personal factors refer to socio-economic conditions, health status, involvement/commitment, adaptation to the living environment, as well as motivation and personal resources. Environmental factors refer to the accessibility of activities (means of transport), existing socialization spaces, participation adaptations related to physical limitations, knowledge of existing activities, place of residence (rural/urban) (Brynjolfsdottir, Palmadottir, & Arnadottir., 2021), or the possibility of carrying out activities outside the place of residence. These factors have also been observed in homes for the elderly. In this respect, geographical location and the quality of communal and private spaces are recognized as factors that sometimes facilitate, sometimes hinder, PS



(Kemp, Ball and Perkins., 2012). The social environment is also identified in studies relating to specialized living environments for seniors, notably the quality and stability of care staff in residences/institutions, geographical location and the quality of relationships with the entourage (Andrianova & Raymond, 2021). Finally, factors related to social networks highlight the influence of a social circle (formal, informal, cultural) pre-existing old age. In addition to these "objective" factors, subjective factors can be added, linking them to personal factors. Thus, PS "responses to obstacles" such as minimizing difficulties or withdrawing into solitary activities, social fears (e.g. rejection, judgment) and the fear of losing preferred identities (Goll et al., 2015) constitute obstacles to PS linked to the question of identity applicable to the older person. From this observation stems a need to consider these determinants in a non-isolated way, taking into account the interactions between them (Townsend, Chen and Wuthrich., 2021). In particular, some authors have observed a relationship between environmental factors, personal factors and SP (Nielson, Wiles and Anderson, 2019; Raymond & Lacroix, 2016). For example, certain characteristics such as motivation and resilience would modulate barriers to participation. However, there are very few studies establishing relationships between the various determinants. Moreover, it seems that these determinants are not fixed; depending on circumstances, facilitators of PS can become obstacles to it, and vice versa. A contingent approach to these determinants is therefore essential if we are to understand the levers of social participation. The literature also notes that it is impossible to generalize results, or even to "establish a recipe for social participation" in retirement homes (Andrianova & Raymond, 2021). There is therefore no predictable, transferable model of social participation.

Sense of community belonging and social participation: At the same time, a sense of belonging and social cohesion are prerequisites both for the health (Cramm & Nieboer, 2015; Valle Panter, 2013) of older people and for social participation (Carver et al., 2018). Indeed, in this study, inclusion in a community, the availability of social resources and the quality of relationships between neighbors within a neighborhood, within a city, would influence and prevent, where appropriate, the frailty of the elderly. Seniors would also be less isolated. In other words, where you live plays a key role in social relations (Bonifas et al., 2014).

Specificity of living environments: In a residential context, the desired "community" context questions the conditions for creating this sense of belonging. Certain structures built around social identity are thus appearing today, such as Alzheimer's homes and "villages" (Cucchi, 2017, 2019; Gentile, 2020), or retirement homes addressed to a population sharing similar characteristics, such as deafness, to offer a living environment that meets specific needs (Hiddinga & Olivier, 2018). In non-institutionalized residential settings, the question of social participation is also raised in view of the desire to offer "a ready-made community for residents who want an inclusive and socially engaged lifestyle". Indeed, the principle of community is not without influence on the quality of life of the elderly (Évans, 2009). Alongside the creation of environments conducive to PS, it would seem that the quality of social relationships (positive, meaningful, reciprocal) is essential in these specific spaces, in order to preserve the psychological health of seniors. Involvement and activities are ways of creating contact with other residents, right from the moment seniors arrive in a new living environment. Group ties are particularly significant, if not more so than individual ties (Haslam et al., 2016); in this sense, shared social identity sometimes plays a major role in the latter (Le Guen, 2001). As the individual factor affects participation, social engagement is not automatic (Park et al., 2010). What's more, the offer is not always easy to apply.

Methodologies used: The elderly person is at the heart of this study, and must be the main actor. Among the intervention typologies and evaluations, the studies insist on this point in order to gain the support of the people involved. The studies surveyed seem to have adopted a research methodology centred on the individual, with an individualized approach, choosing to conduct semi-directive interviews in the case of qualitative studies. There appear to be few studies using a methodology incorporating group interviews

#### Research objectives

Aim of the study: The aim of our study is to propose a model of social participation that emphasizes the creation of a community spirit, and that can be transferred from one residence to another with our partner.

By adopting a contingent approach, we hope to visit several residences with different characteristics, in order to identify the challenges and levers of social participation, as well as their interactions. In addition, we want to understand the



conditions under which a community spirit can be effectively federated and implemented, while at the same time marking out and preventing the possible drifts of an exacerbated communitarian spirit. Our study is intended to be participatory. Through a co-construction approach (Living Lab) that places the elderly person at the heart of our approach, we want the elderly person to feel that they are an actor in their own reality, so as to create conditions that will ensure the long-term benefits of the project.

General objective: To propose a model of social participation that fosters a sense of community among seniors, and that can be transferred to Groupe Maurice residences

# Specific objectives:

- a. Explore and understand the facilitators and challenges of social participation in a residential setting
- b. Explore and understand the facilitators and challenges of creating a sense of community in a residential setting
- c. Test the feasibility of the model
- d. Assess the transferability of the model.

#### RESEARCH METHODOLOGY

#### Research location

Participants and caregivers working in partner settings will not have to travel to TOPMED's premises to take part in data collection (questionnaires, individual interviews, group discussions). Members of the research team will travel to participants' living and/or care environments to conduct the sessions.

For Le Groupe Maurice, two residences co-determined with the partner are included: Gibraltar and Ékla.

All data will be analyzed on TOPMED's premises at 755 Grande-Allée Ouest, Collège Mérici, Quebec City.

# Measurement, assessment and data collection instruments

The study is a living-Lab action-research project.

One of the special features of this research is the implementation of a project support group: this group acts in a consultative capacity, with the role of carrying out operational monitoring of the project (progress of tasks, reporting of unforeseen events and difficulties for each research cycle). There will be 7 meetings, with 6 to 8 volunteer members representing the diversity of residents (new resident, former resident, with and without functional limitations, male, female, caregiver). They will be invited to comment on the project if they have any, and may ask questions if they wish. Meeting minutes will be taken for follow-up purposes, and comments will be audio-recorded and transcribed by the research team. These comments will be used to improve the operational progress of the project

Exchanges will be audio-recorded.

#### Action research cycle 1

The first cycle of action research will establish a realistic picture of social participation and community spirit in two residences co-determined with the partner.

It will be carried out with residents of the targeted residences. It involves a combination of questionnaires and individual interviews

On a voluntary basis, residents will be invited to complete a 20-minute, 10-item paper or digital questionnaire to collect the following data

Socio-demographic data;



- Sense of belonging to a group
- Influence
- Emotional bond

A questionnaire will also be sent to the residence's employees. This questionnaire will focus on their perception of the presence of a community spirit and a sense of belonging on the part of residents.

The following data will be collected:

- Socio-demographic data;
- Sense of belonging to a group
- Influence
- Emotional bond

At the same time, individual 60-minute face-to-face or telephone interviews will be conducted with residents to gather their perceptions of community spirit in the partner's two target residences. The interview guide will cover the following points:

- The concepts of community spirit and sense of belonging
- Facilitating factors
- Obstacle factors
- Existing resources

Interviews can be conducted face-to-face or remotely (via telephone or Teams platform). Interviews will be audio-recorded to facilitate data analysis.

Deliverable: Portrait of community spirit and social participation in each residence

During the project presentation, volunteer participants will be invited to give their opinion on the portrait presented. This will be followed by a 15-minute exercise to formulate a common definition of community spirit. Comments will be audiovideo recorded to facilitate data collection.

# **Estimated duration of participation**

Project support group: Total duration (240 minutes: 1 meeting of 60 minutes and 6 meetings of 30 minutes)

The meetings will be detailed as follows:

- Meeting 1: Reading and signing of FIC (if applicable) (15 minutes)
- Meeting 1-2-3-4-5-6-7: Follow-up on the operational progress of the project and answer questions and gather feedback. (30 minutes)

Action research cycle 1: Total duration (140 minutes)

- Resident questionnaire: (20 minutes)
- Individual resident interview: (60 minutes)
  - Reading of the FIC and signature if applicable (15 minutes)
  - Completion of socio-demographic form (5 minutes)
  - Interview guide (40 minutes)
- Manager questionnaire: (15 minutes)
- Presentation of results: (60 minutes)



- FIC reminder: (10 minutes)

- Results: (20 minutes)

Reflective exercise-defining community spirit (10 minutes)

Gathering comments: (15 minutes)

#### SCIENTIFIC JUSTIFICATION FOR USING LIVE SUBJECTS

The participation of living human subjects representative of the clientele is essential for the collection of data that will enable the creation of user guides adapted to the reality of seniors. The collection of observable and measurable data on the determinants of community spirit will enable us to mobilize seniors to encourage social participation. Data collection will also help us to understand the potential levers for establishing a community spirit in the collective living environment on a long-term basis. It would be impossible to validate these data without living subjects.

#### PARTICIPATION OF SUBJECTS

In each residence co-determined with the partner, we aim to recruit: 50 independent resident volunteers and 5 facility manager volunteers. Here are the details for the project support group and each feedback loop:

- Project support group: 6 to 8 residents
- Research cycle 1: 20 residents for questionnaires and individual interviews; 5 staff members for questionnaires

#### Inclusion criteria:

For Groupe Maurice managers

- Management at Groupe Maurice's Ékla and Gibraltar residences
- Head of department

or

Hold a General Manager position

or

• Be a member of the Groupe Maurice head office

#### For residents

- Residents of the independent wing of Groupe Maurice's Ekla and Gibraltar residences
- Caregiver of a resident of the residences included in the research project

#### **Exclusion criteria:**

For Groupe Maurice staff and residents

- Neurocognitive disorders
- Significant language difficulties
- Lack of verbal communication

#### RECRUITMENT

#### Suitable persons

<u>Managers</u>: Recruitment information on the research project will be distributed in the employee break room. Those interested will be invited to submit their names to the research team via the studies site, topmed. The research team will then send them an e-mail containing a link to an information and consent form. The information and consent forms will be available in digital format at least two weeks before our first visit. During this period, a member of the research team will remain available to answer any questions



Residents of the independent wing: Information about the research project will be disseminated via the Maurice group's internal communication media, which will be co-determined with them. In addition, posters will be distributed to residents' mailboxes. Research activities will be integrated into the residences' calendar in agreement with Groupe Maurice. On a voluntary basis, participants will be able to contact the Topmed research team in order to participate in the various data collection activities, or to express their interest in participating at the residence reception desk and pick up consent forms at the residence reception desk or in the Leisure Manager's office. A period of two (2) weeks will be allowed for reading and reflection. At each meeting, participants will be reminded of the consent form and asked to revalidate their participation. Research activities will then take place.

#### MEASURES AND STRATEGIES TO PROTECT VULNERABLE OR DEPENDENT PERSONS

In this project, participants are recruited on a voluntary basis (stakeholders and residents). Given the project's focus on discussion and exchange on community spirit, good verbal communication and analytical thinking skills are required. Some seniors who find it more difficult to communicate may be accompanied by their caregivers. For people in dependency situations as well as employees, the latter will be recruited on a voluntary basis with a specific procedure ensuring accessibility and signature of online consent forms. Participation will be online or in groups of similar hierarchical level, to ensure freedom of expression and avoid the possibility of undue influence in study participation

#### RISKS AND DRAWBACKS, AND PROPOSED MITIGATION MEASURES

#### Disadvantages:

For managers

The length of time it takes to complete the questionnaire and participate in the results-sharing sessions may
entail some inconvenience, such as a slight disruption to work schedules and daily tasks. Meetings will be
scheduled in agreement with the partner environment.

#### For residents

This project may entail some inconvenience, such as a slight disruption to the schedule of activities and the
possibility of emotional reactions. Wherever possible and appropriate, research activities will be planned and
confirmed in advance.

# **Risks**

# Questionnaire

There is no risk associated with completing the guestionnaire.

#### Individual interviews

As far as we are aware, apart from the time spent on the interview, participation in this study will not cause
any physical or psychological harm to the participant. However, it remains possible that the discussion of
certain themes may make the participant uncomfortable or give rise to discomfort. In such cases, participants
are free not to answer certain questions. If necessary, they can be referred to appropriate support resources.

#### Focus groups, working groups and prioritization workshops

As far as we know, apart from the time spent on the interview, participation in this study will not cause any
physical or psychological harm to the participant. However, it remains possible that the discussion of certain
themes may make the participant uncomfortable or give rise to discomfort. In such cases, participants are free
not to answer certain questions. If necessary, they can be referred to appropriate support resources.



Despite the means put in place to ensure the confidentiality of group discussions, certain risks inherent in this
type of consultation cannot be avoided. In other words, the research team cannot guarantee that each group
participant will keep the information exchanged confidential

#### Process

- Participation difficulties: the person may fear being judged or rejected. The research team will ensure that conditions are in place to create a safe space for expression, including a climate of emotional security
- There may be variations in the person's state of health (fatigue, age-related cognitive loss) or difficulties
  getting around. The research team will make sure to establish consultation times that respect the person's
  health conditions, by choosing discussion areas that are accessible to all.
- Have only socially active people participate in the project. The research team will make sure to reach all residents for recruitment and allow participants to choose their participation formula: individual or group.
- Difficulty in keeping people actively involved over the medium-to-long term (the project period): people
  withdraw while the study is being carried out, and may lose the sense of their participation. Explain the
  project's objectives, and monitor progress from one session to the next, to encourage buy-in and commitment.
  Put the individual at the heart of the project: the individual level must be present in the approach and
  discussions, so that participants can find meaning in their participation each time.

#### **ADVANTAGES AND BENEFITS**

Benefits for partner managers

It is anticipated that the research project will support community spirit within the observed environment, as well as the possibility of implementing the concept in all the partner's residences.

#### Benefits for senior participants

We expect to see an increase in the active social participation of seniors. In addition, this project will provide an opportunity to reflect on solutions that will enable seniors to evolve in an environment that resembles their own, and that favors the inclusion of everyone, thus combating isolation

#### Project benefits

The participation of seniors will enable us to better target the needs of different environments, and gather data on the facilitating factors and challenges of community spirit and social participation. The participation of seniors will enable us to better target their needs and interests in order to develop solutions adapted to the clientele.

#### FREE AND INFORMED CONSENT

The information and consent form will be available online (for staff) and in hard copy (for residents) at two locations in the partner community (reception and recreation manager's office). Participants will be able to obtain a copy of the document to familiarize themselves with its contents. A two-week period for reading and reflection will be given staff and resident participants. During this time, they will be able to contact a member of the research team for further information or to ask questions about the project and its progress, if applicable. Completed FICs can be handed in at the reception desk or at the leisure leader's office, in a sealed envelope. During the meetings, the form will be reexplained and the potential participant will be free to consent to take part in the research project. At any time, the participant may decide to end his or her participation.

For the possibility of meeting people on the Teams platform, an explicit registration consent request will be set up.

# CONFIDENTIALITY AND PROTECTION OF PERSONAL INFORMATION

The ethics committee that evaluated the project can access the research data for control and verification purposes



All information collected will remain strictly confidential to the extent permitted by law. In order to preserve the identity of participants and the confidentiality of information, participants will be identified by a code. The list of codes linking a name to a research file will be kept in the office of the responsible researcher, in a locked filing cabinet at TOPMED at Mérici Collégial Privé, 755 Grande Allée Ouest, Québec, Qc, G1S 1C1. Unless required by law, no information that could directly or indirectly reveal the identity of subjects will be released or published without their prior explicit consent.

As part of the project, consent forms presented in digital form are created using the Lime Survey platform. The information processed is hosted in Canada on the platform's encrypted servers (Secure Socket Layer procedure), which comply with the RGPD standard. In addition, participants will not be required to consent to the platform's terms and conditions

Regarding the methods of storing and securing audio-video recordings, these will be made by cameras recording the data on SD cards. Video captures are confidential and will only be used for the purposes of this research project, unless otherwise agreed by the participant or his/her legal representative. All data collected will be encrypted on servers. Unless required by law, no information that could directly or indirectly reveal their identity will be distributed or published without their prior explicit consent. Only members of the research team (all subject to confidentiality) will have access to participants' identifying information and encrypted research data, which will be kept separate from research materials, data and information and consent forms.

Documents will be kept for a period of five (5) years following collection, after which they will be destroyed. During this 5-year retention period, if data is stored on a USB key or other external medium, it will be encrypted.

Any scientific publication resulting from this research project will present statistical data only, and under no circumstances will the names of the participants be published or divulged to anyone.

#### **CONTINUOUS EXAMINATION**

Should any inconvenience arise during project validation, subjects will be promptly notified.

#### **DISSEMINATING RESULTS**

No disclosure to participants will be made following completion of their participation.

#### **COMPENSATION**

Stakeholders receive no financial compensation for their participation in the research project.

For residents, there is financial compensation for participation in the research project.

However, for each activity, if no monetary remuneration is given, we will offer snacks to participants following the sessions.

#### RESPONSIBILITY

The legal rights of each subject will be maintained.

#### CONFLICT OF INTEREST AND PROPOSED MITIGATION MEASURES

No conflict of interest.

#### PROTOCOL SEQUENCE

# **Posters**

437\_Affich-Recrut-site\_études Posters-social participation-recruitment-V2



# **Admission**

437\_Email\_Recruit

# **Project support group**

437\_FIC\_Project\_Support\_Group

# First research cycle

# Consent form

- 437\_FIC\_Residents\_Cycle 1
- 437\_FIC\_Management\_Cycle 1-2-3
- 437\_FIC\_Presentation\_Results Cycle 1-2-3

# Measuring instruments

- 437\_Individual interview guide
- 437\_Questionnaire\_Residents\_GM
- LimeSurvey Cloud Your online survey service 437\_Questionnaire\_EspCom\_Gestion

# **Data processing**

Compilation of questionnaires, interviews, prioritization workshops and results presentation sessions

#### **Compilation of**

Data analysis without statistical inference tests